CLINICAL TRIAL: NCT00499655
Title: A Randomized, Placebo-Controlled Phase II Clinical Trial of Combination Erlotinib (Tarceva) and Celecoxib (Celebrex) Versus Erlotinib (Tarceva)/Placebo in Advanced Non-Small Cell Lung Cancer Patients
Brief Title: Erlotinib Hydrochloride With or Without Celecoxib in Treating Patients With Stage IIIB-IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06254; NCI-2010-00353 (Registry Identifier: NCI CTRP); CDR0000549751 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Celecoxib; Immunohistochemistry; In Situ Hybridization, Fluorescence; Gene Expression Profiling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oral erlotinib hydrochloride once daily and oral placebo twice daily on days 1-28.
  Interventions: Drug: erlotinib hydrochloride; Other: placebo; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: fluorescence in situ hybridization; Genetic: mutation analysis; Genetic: protein expression analysis; Genetic: gene expression analysis
- Arm II (Experimental): Patients receive oral erlotinib hydrochloride once daily and oral celecoxib twice daily on days 1-28.
  Interventions: Drug: erlotinib hydrochloride; Drug: celecoxib; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: fluorescence in situ hybridization; Genetic: mutation analysis; Genetic: protein expression analysis; Genetic: gene expression analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774; Tarceva
Drug: celecoxib — Given orally
  Other Names: Celebrex; SC-58635; YM 177
  Arms: Arm II
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Genetic: mutation analysis — Correlative studies
Genetic: protein expression analysis — Correlative studies
Genetic: gene expression analysis — Correlative studies

SUMMARY:
RATIONALE: Erlotinib hydrochloride and celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Celecoxib may also stop the growth of lung cancer by blocking blood flow to the tumor. Giving erlotinib hydrochloride together with celecoxib may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving erlotinib hydrochloride together with celecoxib works compared with erlotinib hydrochloride alone in treating patients with stage IIIB-IV non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Comparison of progression-free survival (PFS) in patients receiving erlotinib + celecoxib vs. erlotinib + placebo for advanced NSCLC.

SECONDARY OBJECTIVES:

I. Objective tumor response rate as defined by RECIST Criteria for subjects receiving erlotinib/celecoxib treatment arms.

II. Categorize the change in e-cadherin expression from baseline to week 8 in a subset of subjects.

III. Evaluation of overall survival (OS). IV. Measurement of COX-2, EGFR by immunohistochemistry and EGFR amplification by FISH, and EGFR mutation status to correlate with clinical response.

V. Measurement of change in urinary PGE-M and correlation with response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral erlotinib hydrochloride once daily and oral placebo twice daily on days 1-28.

ARM II: Patients receive oral erlotinib hydrochloride once daily and oral celecoxib twice daily on days 1-28.

In both arms, treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* Pathologically proven NSCLC, stage IIIB (defined as: with pleural effusion or recurrence after mediastinal radiation and chemotherapy) or IV
* Available tumor tissue for mutation screening
* Measurable stage IIIb or IV disease by RECIST guidelines
* ECOG performance status of 0 or 1
* Progressive disease despite >= 1 prior chemotherapy regimens as standard of care or subject's refusal or inability to receive standard chemotherapy
* Normal renal function (defined as serum creatinine =< 2mg/dl)
* Normal liver function (defined as serum total bilirubin =< 1.5, and serum transaminases =< 2.5X the upper limits of normal [ULN]); if liver metastases are present, serum transaminases > 5X the ULN
* No evidence of coagulopathy (defined as PT and/or PTT =< 1.5X ULN or platelets >= 100,000)
* No evidence of leukopenia (defined as absolute neutrophil count >= 1,500 mm^3)
* Negative pregnancy test prior to initiation of treatment and adequate contraception throughout treatment

Exclusion

* Cytotoxic chemotherapy agents within 4 weeks of initiating treatment; all toxicities must be recovered to baseline or NCI CTCAE v3.0 Grade 1 from all acute effects of prior cancer treatment, except alopecia or any clinically insignificant effect, prior to study initiation
* Evidence of NYHA class III or greater cardiac disease, history of myocardial infarction, cerebral vascular accident, symptomatic ventricular arrhythmia, or symptomatic conduction abnormality
* Non-cytoxic therapy within 2 weeks of initiating treatment ; all toxicities must be recovered to baseline or NCI CTCAE v3.0 Grade 1 from all acute effects of prior cancer treatment, except alopecia or any clinically insignificant effect, prior to study initiation
* Prior radiotherapy to target lesions is not permitted unless completed more than 4 weeks prior to treatment within the study and that there has been documented progression at these sites (Radiotherapy to non-target lesions is permitted within 2 weeks of study entry provided all acute effects of the radiotherapy have resolved at least grade 1)
* Comorbid disease or a medical condition that would impair the ability of the subject to receive or comply with the study protocol
* Prior malignancy within the last 3 years with the exception of non-melanoma skin cancer or cervical cancer in situ
* Hypersensitivity of erlotinib or celecoxib or to any of the excipients of these products
* Hypersensitivity to sulfonamides, aspirin or other NSAIDS
* Prior history of EGFR inhibitor for the treatment of cancer
* Previous history of gastrointestinal ulceration, bleeding or perforation
* Concurrent use of COX-2 inhibitors or other NSAIDS (For subjects on NSAIDS prior to study initiation, cessation of the drug for 72 hours prior to study entry is required)
* Chronic or concurrent use of steroids (topical steroids are acceptable if medically indicated)
* Subjects who require treatment with fluconazole or lithium
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded)
* Renal insufficiency (defined as serum creatinine > 2 mg/dl)
* Liver insufficiency (defined as serum total bilirubin > 1.5, or serum transaminases > 2.5C the upper limits of normal [ULN]); if liver metastases are present, serum transaminases > 5X the ULN
* Coagulopathy (defined as PT and/or PTT > 1.5X ULN or platelets < 100,000)
* Leukopenia (defined as absolute neutrophil count < 1,500/mm^3)
* Pregnancy or inadequate contraception
* Lactating females
* Active CNS metastasis (stable, treated CNS metastasis acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Reckamp, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib\Placebo: Patients receive 150 mg of oral erlotinib hydrochloride once daily and oral placebo twice daily on days 1-28.
  erlotinib hydrochloride: Given orally
  placebo: Given orally
  laboratory biomarker analysis: Correlative studies
  immunohistochemistry staining method: Correlative studies
  fluorescence in situ hybridization: Correlative studies
  mutation analysis: Correlative studies
  protein expression analysis: Correlative studies
  gene expression analysis: Correlative studies
- Erlotinib\Celecoxib: Patients receive 150 mg of oral erlotinib hydrochloride once daily and 600 mg of oral celecoxib twice daily on days 1-28.
  erlotinib hydrochloride: Given orally
  celecoxib: Given orally
  laboratory biomarker analysis: Correlative studies
  immunohistochemistry staining method: Correlative studies
  fluorescence in situ hybridization: Correlative studies
  mutation analysis: Correlative studies
  protein expression analysis: Correlative studies
  gene expression analysis: Correlative studies
Period: Overall Study
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Started | 53 | 54
Completed | 53 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Continuous [Median (Full Range); unit: years] | 65 [30 to 80] | 63.5 [41 to 80] | 64 [30 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 24 | 26 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 54 | 107

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST), as a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Until disease progression, up to 5 years.
Population: All patients receiving treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Number analyzed (Participants) | 53 | 54
Months | 3.5 [1.8 to 5.5] | 5.4 [2 to 7.6]

2. Secondary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 16 weeks post start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Number analyzed (Participants) | 53 | 54
Participants | 17 | 12

3. Secondary Outcome: Progression-free Survival - Elevated PGEM
Description: as for outcome 1
Time Frame: Until disease progression, up to 5 years.
Population: Analysis on a subset of patients with elevated baseline urinary prostaglandin E metabolite (PGEM).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Number analyzed (Participants) | 30 | 30
Months | 2.2 [1.8 to 5.5] | 5.4 [1.8 to 12.9]

4. Secondary Outcome: Progression-free Survival - EGRF
Description: as for outcome 1
Time Frame: Until disease progression, up to 5 years.
Population: Analysis on a subset of patients with wild-type epidermal growth factor receptor (EGFR),
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Number analyzed (Participants) | 27 | 31
Months | 1.8 [1.7 to 3.5] | 3.2 [1.7 to 6.7]

5. Secondary Outcome: Progression-free Survival - Low PGEM
Description: as for outcome 1
Time Frame: Until disease progression, up to 5 years.
Population: Analysis on a subset of patients with low baseline urinary prostaglandin E metabolite (PGEM).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Erlotinib\Celecoxib: Patients receive 150 mg oforal erlotinib hydrochloride once daily and 600 mg of oral celecoxib twice daily on days 1-28.
  erlotinib hydrochloride: Given orally
  celecoxib: Given orally
  laboratory biomarker analysis: Correlative studies
  immunohistochemistry staining method: Correlative studies
  fluorescence in situ hybridization: Correlative studies
  mutation analysis: Correlative studies
  protein expression analysis: Correlative studies
  gene expression analysis: Correlative studies
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Number analyzed (Participants) | 15 | 14
Months | 5.4 [1.7 to 7.2] | 6.8 [1.7 to 9.0]

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 6 years.
Arm/Group | Erlotinib\Placebo | Erlotinib\Celecoxib
Serious Adverse Events (participants affected / at risk) | 1/53 | 2/54
Other Adverse Events (participants affected / at risk) | 53/53 | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib\Placebo (N=53) | Erlotinib\Celecoxib (N=54)
cerebrovascular ischemia (Vascular disorders) | 0 (0) | 2 (2)
cardiac ischemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib\Placebo (N=53) | Erlotinib\Celecoxib (N=54)
Rash (Skin and subcutaneous tissue disorders) | 42 (42) | 43 (43)
Diarrhea (Gastrointestinal disorders) | 40 (40) | 38 (38)
Dry skin (Skin and subcutaneous tissue disorders) | 40 (40) | 36 (36)
Fatigue (General disorders) | 31 (31) | 28 (28)
Elevated AST (Investigations) | 27 (27) | 25 (25)
Anorexia (Psychiatric disorders) | 26 (26) | 17 (17)
Nausea (General disorders) | 17 (17) | 14 (14)
Hypoalbuminemia (Investigations) | 14 (14) | 16 (16)
Stomatitis (General disorders) | 12 (12) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 18 (18)
Elevated creatinine (Investigations) | 8 (8) | 17 (17)
Elevated Alk Phos (Investigations) | 11 (11) | 12 (12)
Paronychia (Infections and infestations) | 7 (7) | 16 (16)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 10 (10)
Weight Loss (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Vomiting (General disorders) | 7 (7) | 4 (4)
Elevated bilirubin (Investigations) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes